CLINICAL TRIAL: NCT00050141
Title: A Randomised, Blinded, Phase 2 Study of Letrozole Plus the Farnesyl Transferase Inhibitor ZARNESTRA TM (R115777) and Letrozole Plus Placebo in the Treatment of Advanced Breast Cancer After Antiestrogen Therapy.
Brief Title: Study of Letrozole Plus Tipifarnib or Placebo in the Treatment of Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004030; NCT00060177 (obsolete NCT alias); NCT00723372 (obsolete NCT alias)
Record Dates: First submitted 2002-11-22; First posted 2002-11-28 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Breast Cancer
Keywords: Breast cancer; ZARNESTRA; tipifarnib; R115777; Estrogen receptor positive; Progesterone receptor positive; Anti-estrogen therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — tipifarnib

INTERVENTIONS:
Drug: ZARNESTRA, tipifarnib, R115777

SUMMARY:
The purpose of this study is to determine if the addition of tipifarnib to standard letrozole therapy leads to a better response to treatment for your cancer in comparison to letrozole plus a placebo. Tipifarnib belongs to a class of drugs called Farnesyl Transferase Inhibitors (FTI). It blocks proteins that make cancer cells grow.

DETAILED DESCRIPTION:
This clinical study involves two groups of patients with advanced breast cancer. One group (2/3rds of all the patients) will be taking tipifarnib in combination with another anticancer drug called letrozole, and the other group (1/3rd of all the patients) will be taking letrozole plus a placebo (an inactive substance given in the same form as a real drug). The assignment to one of these two groups will be by chance (like flipping a coin). Unless the need arises, neither the patient nor the study staff will know whether the patient is receiving tipifarnib with the letrozole. Comparisons between the two groups will be made for patients who have achieve a confirmed Complete Response (CR) or Partial Response (PR). The interval between the date of randomization and the earliest date of disease progression will also be assessed. The study will include evaluations of safety and tolerability. Patients should expect their participation in this trial to last a minimum of 4 to 8 weeks. Their participation could continue for several months or beyond a year, depending on how their disease responds to the treatment. After completing study treatment, patients will be asked to attend for an End of Treatment visit and then a posttreatment Follow-up visit 4 to 6 weeks after stopping the medication. Patients will be randomly assigned to treatment with either 2.5 mg letrozole once daily plus placebo to match tipifarnib twice daily, or 2.5 mg letrozole once daily plus 300 mg tipifarnib twice daily. Both tipifranib and matching placebo will be given in 28-day cycles of 21 days of treatment followed by 7 days rest. All patients will receive continuous treatment with letrozole.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced, inoperable loco-regionally-recurrent, or metastatic breast cancer
* Estrogen and/or progesterone positive disease
* Progression of disease after antiestrogen therapy
* Measurable disease
* Postmenopausal
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2.

Exclusion Criteria:

* Previous endocrine therapy, other than antiestrogen therapy
* More than 1 prior chemotherapy regimen
* Previous therapy with farnesyl transferase inhibitor
* Presence of rapidly progressive, life-threatening metastases
* Concomitant anticancer treatment
* Other malignancy within the past 5 years
* Symptomatic peripheral neuropathy.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2002-09; Primary Completion 2005-10 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Comparisons between the two treatment groups will be made for patients who have achieve a confirmed Complete Response (CR) or Partial Response (PR).

SECONDARY OUTCOMES:
Effectiveness will be assessed by time to disease progression; time to treatment failure; duration of response; clinical benefit; duration of clinical benefit; survival time. The study will include evaluations of safety and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (23):
- United States (6):
  - Miami, Florida
  - Chicago, Illinois
  - Durham, North Carolina
  - Cleveland, Ohio
  - Fort Worth, Texas
  - Tyler, Texas
- Belgium (2):
  - Brussels
  - Leuven
- France (6):
  - Bordeaux
  - Clermont-Ferrand
  - Montpellier Cedex 5 N/A
  - Rennes
  - Saint-Herblain
  - Vandœuvre-lès-Nancy
- The Hague, Netherlands
- Russia (2):
  - Moscow
  - Saint Petersburg
- United Kingdom (6):
  - Huddersfield
  - Leeds
  - London
  - Manchester
  - Newcastle upon Tyne
  - Sutton

REFERENCES:
- [Derived] Johnston SR, Semiglazov VF, Manikhas GM, Spaeth D, Romieu G, Dodwell DJ, Wardley AM, Neven P, Bessems A, Park YC, De Porre PM, Perez Ruixo JJ, Howes AJ. A phase II, randomized, blinded study of the farnesyltransferase inhibitor tipifarnib combined with letrozole in the treatment of advanced breast cancer after antiestrogen therapy. Breast Cancer Res Treat. 2008 Jul;110(2):327-35. doi: 10.1007/s10549-007-9726-1. Epub 2007 Sep 13. PMID 17851757
- See also: Pharmacoepidemiologic International Longitudinal Antipsychotic Registry PILAR — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=397&filename=CR014707_CSR.pdf